CLINICAL TRIAL: NCT00618215
Title: Impact of Multifaceted Peer Group Education to Improve Routine Oral Examinations in Primary Care A Cluster-Randomised Controlled Trial
Brief Title: A Cluster Randomized Controlled Trial in Primary Oral Care
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: The health Care Insurance Board (CVZ) (Unknown); Department of Preventive and Restorative Dentsitry and Centre of Quality of Care Research (WOK) (Unknown)
Responsible Party: Prof. dr. A. Plasschaert, Prof. dr R. Grol
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: CVZ-538/001/2001/RL000003
Record Dates: First submitted 2008-02-05; First posted 2008-02-19 (Estimated); Last update posted 2008-02-19 (Estimated); Status verified 2008-02

CONDITIONS: Tooth, Impacted
Keywords: cluster-randomised trial; routine oral examination; implementation research; practice based research; CPG; recall interval assignment for routine oral examination; prescription bitewing radiographs; preventive advice and feed back oral disease
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): ROE Group
  Interventions:behaviorial
  Interventions: Behavioral: peer group educational implementation strategy
- 2 (Experimental): MIM Group
  Interventions:behaviorial
  Interventions: Behavioral: peer group educational implementation strategy

INTERVENTIONS:
Behavioral: peer group educational implementation strategy — Delivery CPG
  Education session IQual group
  Online training website (individual feed back)
  Reminder (flow chart), individual feed back record form
  Feed back by email
  Registration in practice

SUMMARY:
Background: Routine oral examination (ROE) refers to periodic monitoring of the general and oral health status of patients. In most developed Western countries a decreasing prevalence of oral diseases underpins the need for a more individualised approach in assigning recall intervals for regular attendees instead of systematic decision making of fixed intervals. From a quality of care perspective as well, one can also question the effectiveness of the widespread prophylactic removal of mandibular impacted asymptomatic third molars (MIM) in adolescents and adults. It is as yet unclear how quality of oral care can be improved. Research data on effectiveness of interventions to promote continuing professional development for dentists are rare.

Methods/Design: This implementation study is a cluster randomised controlled trial with groups of GDPs as the unit of randomisation. The aim of the study is to determine the effectiveness and efficiency of small group quality improvement on professional decision making of general dental practitioners (GDPs) in daily practice. Six peer groups ('IQual-groups') shall be randomised either to the intervention group I or group II. Groups of GDPs allocated to either of these arms act as each other's control group. An IQual peer group consists of 8-10 GDPs who attend in monthly structured sessions scheduled for discussion on practice related topics.

GDPs in both trail arms receive recent developed evidence-based CPG on ROE or MIM respectively. The implementation strategy consists of 1 interactive IQual circle meeting of mostly 2-3 hours. In addition, both groups of GDPs receive feedback on personal and group characteristics and are invited to make use of web-based patient vignettes for further individual training on risk assessment policy. A few weeks after the interactive meeting reminders (flow charts) will be send by mail.

The main outcome measure for the ROE-study and control group is the use and appropriateness of individualised risk assessment in assigning recall intervals and for the MIM-study the use and appropriateness of individualised mandibular impacted third molar risk management.

Measurements (pre-intervention data collection) will take place in months 1-3, starting in September 2006. Post-intervention data collection will be performed after 9 months.

Discussion: In most developed Western countries a decreasing prevalence of oral diseases underpins the need for a more individualised approach in assigning recall intervals for regular attendees. If the evaluation of this multifaceted implementation study reveals a shift in individual performance of GDPs in assessing risks for oral disease, further research questions and efforts to a risk-based professional education could be promoted.

Scientific hypothesis Multifaceted implementation of consensus based clinical practice guidelines (CPGs) for GDPs on ROEs and the management of asymptomatic impacted third molars (MIM) in daily dental practice is more effective and efficient compared to only dissemination of CPGs.

ELIGIBILITY:
Inclusion Criteria:

GDPs inclusion criteria

* GDPs have to work in general dental practice for at least three days/week and should have practice experience for at least three years. They were eligible if their practice population was characterised by primary oral care patients, consisting of regular attendees, and patient recordkeeping was conducted electronically. GDPs had to give their informed consent to assess and evaluate electronically patient records. Patient data were collected anonymously.

Patient's inclusion criteria

To be eligible for inclusion, patients should meet (fulfil) several criteria, depending on the IQual's CPG to be used (ROE or MIM):

ROE:

* All patients regularly visiting their dentist (at least once a year) over the past three years for ROEs will be included in the study.

MIM:

* All patients regularly visiting their dentist (at least once a year) over the past three years for ROEs are included for the study and, in addition, have to be aged between 17 and 35 years, with disease-free impacted mandibular third molars in retention.

For both group of patients, it is important that they can be linked particular to the participating GDP, especially in practices with more than one GDP occupied

Exclusion Criteria:

Patient's exclusion criteria

ROE:

* Patients with symptomatic driven (emergency) attendance in dental practice, or recently started regular attendance in the participating dental practice (within past three years).

MIM:

* Patients with symptomatic third molars in dental practice, or recently started regular attendance (past three years) or who already had their third molars removed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1161 (Actual)
Dates: Start 2006-09; Primary Completion 2007-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Number of patients per GDP with assigned recall interval (months) based on individual recall assessment. For high risk children and adolescents <7 months, in case of low risk > 7 months. For adults 9 months or more for low risk profiles, and ≤ than 9 mo | September 2006 and June 2007

SECONDARY OUTCOMES:
Number of patients per GDP with prescribed individual frequency of BWs (months). For high-risk children and adolescents <24 months frequency, in low risk profiles >36 months. For high-risk adults < 36 months frequency versus low risk >48 months. | september 2006 and june 2007

CONTACTS AND LOCATIONS:
Overall Officials: Alphons Plasschaert, Prof Phd, Principal Investigator — University Medical Centre St Radboud Nijmegen The Netherlands; dirk Mettes, DMD, Study Chair — UMC St Radboud Medical Centre Nijmegen The Netherlands
Locations (1):
- University Medical Centre St Radboud, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Mettes TG, van der Sanden WJ, Wensing M, Grol RP, Plasschaert AJ. A cluster randomised controlled trial in primary dental care based intervention to improve professional performance on routine oral examinations and the management of asymptomatic impacted third molars: study protocol. Implement Sci. 2007 Apr 20;2:12. doi: 10.1186/1748-5908-2-12. PMID 17448224